CLINICAL TRIAL: NCT01093417
Title: The Effect of Vitamin D Supplementation on Endothelial Function, Inflammation and Insulin Resistance in HIV
Brief Title: Study of Vitamin D and Effect on Heart Disease and Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Grace McComsey, Chief, Peds ID, Rheumatology and Global Health, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 11-09-30
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Human Immunodeficiency Virus (HIV); Vitamin D Deficiency; HIV Infections
Keywords: Vitamin D; Human Immunodeficiency Virus (HIV); Complementary Therapies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Vitamin D Deficiency; HIV Infections | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants that have been randomized into this arm will receive placebo pills.
  Interventions: Other: Placebo
- Vitamin D 4000 IU (Active Comparator): Participants that have been randomized into this arm will receive Vitamin D 4000 IU (International Units) daily.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 4000 IU will be administered to enrollees on the active comparator arm
  Other Names: Calciferol
  Arms: Vitamin D 4000 IU
Other: Placebo — Placebo pills will be administered to enrollees in this arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how Vitamin D affects endothelial function, inflammation, lipids, insulin resistance, vitamin D levels, and parathyroid hormone (PTH).

DETAILED DESCRIPTION:
Randomized placebo controlled trial of vitamin D supplementation in HIV infected subjects with vitamin D deficiency

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* HIV-RNA < 400 copies/ml at study entry and for 12 wks. prior
* 25-hydroxyvitamin D level <20
* On a stable anti-retroviral (ARV) regimen for at least 12 weeks prior to study entry

Exclusion Criteria:

* Pregnancy or Breast Feeding
* Diabetes
* Creatinine Clearance <50
* Any active infectious or inflammatory condition
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 within 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Longenecker CT, Hileman CO, Carman TL, Ross AC, Seydafkan S, Brown TT, Labbato DE, Storer N, Tangpricha V, McComsey GA. Vitamin D supplementation and endothelial function in vitamin D deficient HIV-infected patients: a randomized placebo-controlled trial. Antivir Ther. 2012;17(4):613-21. doi: 10.3851/IMP1983. Epub 2011 Nov 17. PMID 22293363

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 15 participants were randomized to matching placebo for 12 weeks
- Vitamin D 4000 IU: 30 participants were randomized to 4000IU of cholecalciferol (vitamin D3) daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Vitamin D 4000 IU
Started | 15 | 30
Completed | 15 | 29
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D 4000 IU | Total
Number analyzed (Participants) | 15 | 30 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 30 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10) | 47 (8) | 45 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 25 | 35
Region of Enrollment [Number; unit: participants]
  United States | 15 | 30 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelial Function
Description: Endothelial function measured by flow mediated brachial artery dilation
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: percent change in endothelial function
Arm/Group | Placebo | Vitamin D 4000 IU
Number analyzed (Participants) | 15 | 29
percent change in endothelial function | 0.29 [-1.61 to 1.77] | 0.55 [-1.05 to 2.13]

2. Secondary Outcome: Change in Serum 25-hydroxyvitamin D Concentration in Both Groups
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Vitamin D 4000 IU
Number analyzed (Participants) | 15 | 29
ng/mL | -1.8 [-2.9 to 0.1] | 5.0 [-0.9 to 7.4]

ADVERSE EVENTS:
Arm/Group | Placebo | Vitamin D 4000 IU
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/30
Other Adverse Events (participants affected / at risk) | 0/15 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes